CLINICAL TRIAL: NCT06220201
Title: A Phase 1, Multicenter, Single-arm, Dose-escalation Study of CC-97540 (BMS-986353), CD19-Targeted NEX-T Chimeric Antigen Receptor (CAR) T Cells, Evaluating Safety and Tolerability in Participants With Autoimmune Neurological Diseases: Relapsing Forms of Multiple Sclerosis (RMS), Progressive Forms of Multiple Sclerosis (PMS), or Refractory Myasthenia Gravis (MG).
Brief Title: A Study to Evaluate the Safety, Tolerability, Efficacy, and Drug Levels of CC-97540 in Participants With Relapsing Forms of Multiple Sclerosis, Progressive Forms of Multiple Sclerosis or Refractory Myasthenia Gravis (MG) (Breakfree-2)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA061-1006; 2023-507820-22 (Other: EU CT Number); U1111-1296-8579 (Other: UTN)
Record Dates: First submitted 2024-01-04; First posted 2024-01-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis; Myasthenia Gravis
Keywords: CC-97540; CAR T; CART; NEX T; NEXT; BMS-986353; RMS; PMS; Multiple sclerosis; RRMS; aSPMS; PPMS; iSPMS; MG; gMG; refractory myasthenia gravis; general myasthenia gravis; CD19
MeSH Terms: conditions — Multiple Sclerosis; Myasthenia Gravis | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Administration of CC-97540 (RMS arm) (Experimental)
  Interventions: Drug: CC-97540; Drug: Fludarabine; Drug: Cyclophosphamide
- Administration of CC-97540 (PMS arm) (Experimental)
  Interventions: Drug: CC-97540; Drug: Fludarabine; Drug: Cyclophosphamide
- Administration of CC-97540 (MG arm) (Experimental)
  Interventions: Drug: CC-97540; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CC-97540 — Specified dose on specified days
  Other Names: BMS-986353
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, efficacy, and drug levels of CC-97540 in participants with Relapsing Forms of Multiple Sclerosis (RMS), Progressive Forms of Multiple Sclerosis (PMS) or Refractory Myasthenia Gravis (MG).

ELIGIBILITY:
Inclusion Criteria

- Relapsing forms of Multiple Sclerosis (RMS) - Cohort 1.

i) Participants must have an Expanded Disability Status Scale (EDSS) of ≥ 3.0 and ≤ 5.5.

ii) Participants must have a diagnosis of Multiple Sclerosis (MS) with relapsed/refractory MS or conversion to active secondary progressive multiple sclerosis (aSPMS), and worsening of disease within 12 months prior to Screening and while on treatment with a high-efficacy DMT for at least 6 months.

- Progressive forms of MS - Cohort 2.

i) Participants must have an EDSS ≥ 3.0 and ≤ 6.0.

ii) Participants must have a diagnosis of primary progressive multiple sclerosis (PPMS) that is treatment-resistant or diagnosis of inactive secondary progressive multiple sclerosis (iSPMS).

- Myasthenia Gravis - Cohort 3

i)MGFA classification of II-IV at screening

ii) Documentation of autoantibodies against AChR or MuSK (historical or at Screening)

iii) Refractory disease defined as disease activity on at least 2 immunosuppressants, including steroids, NSIs, or biologics.

iv) Has had thymectomy, only if indicated according to current guidelines.

Exclusion Criteria

* Cohorts 1 and 2: Participants that cannot complete the 9-Hole Peg Test (9-HPT) in at least 1 hand in <240 seconds unless extenuating medical conditions unrelated to MS prohibit this.
* Participants that cannot perform a Timed 25-Foot Walk Test (T25FWT) in < 150 seconds.
* Presence of other confounding peripheral nervous system disorders or other disorders that may impact muscle strength (eg, myositis) or cause weakness, stroke, chronic inflammatory demyelinating polyradiculoneuropathy, Lambert-Eaton myasthenic syndrome.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to week 104
Number of participants with serious adverse events (SAEs) | Up to week 104
Number of participants with adverse events of special interest (AESIs) | Up to week 104
Number of participants with laboratory test result abnormalities | Up to week 104
Number of participants with imaging abnormalities | Up to week 104
  For Cohorts 1 and 2
Number of participants with dose-limiting toxicities (DLTs) | Up to week 104
Recommended Phase 2 dose (RP2D) based on the incidence of DLTs that occur during the DLT evaluation period | Up to week 104

SECONDARY OUTCOMES:
Number of participants meeting no evidence of disease activity (NEDA) criteria | Up to week 104
Number of participants with confirmed disability progression per Expanded Disability Status Scale (EDSS) | Up to week 12
Annualized relapse rate | Up to week 104
Change from baseline in magnetic resonance imaging (MRI) metrics | Up to week 104
  MRI metrics assessed are 1) number of gadolinium-enhancing T1 lesions and 2) total number of new or enlarging hyperintense T2-weigted lesions
Number of participants with disability improvement confirmed per EDSS | Up to week 12
Maximum observed blood concentration (Cmax) | Up to week 104
Time of maximum observed blood concentration (Tmax) | Up to week 104
Area under the blood concentration-time curve from time zero to 28 days after dosing (AUC(0-28D)) | Up to week 104
Time to last measurable chimeric antigen receptor (CAR T) concentrations (Tlast) | Up to week 104
Number of participants with at least 2 points improvement for at least 4 weeks in Myasthenia Gravis activities of daily living (MG-ADL) score | Up to week 26
  For Cohort 3
Number of participants with at least 3 point improvement in Myasthenia Gravis composite (MG-C) score | Up to week 26
  For Cohort 3
Number of participants with at least 3 point improvement in quantitative Myasthenia Gravis (QMG) score | Up to week 26
  For Cohort 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Irvine, Irvine, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - University of Kansas Medical Center, Kansas City, Kansas
  - Local Institution - 0039, New Orleans, Louisiana
  - Local Institution - 0005, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Neurological Institute of New York, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Mellen Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - Antwerp University Hospital, Edegem, Antwerpen
  - UZ Gent, Ghent, Oost-Vlaanderen
- France (2):
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
  - Pitie Salpetriere University Hospital, Paris, Ville de Paris
- Germany (5):
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - Local Institution - 0033, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Klinikum der Universität München Großhadern, München
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0016, Barcelona, Barcelona [Barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - Manchester Royal Infirmary, Manchester, Lancashire
  - University College London Hospital, London, London, City of
  - Salford Royal Hospital, Salford, Manchester
  - Barts Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06220201.html